CLINICAL TRIAL: NCT03119493
Title: Effects of Periodized Aerobic Interval Training on Autonomic Modulation and Cardiovascular and Anthropometric Variables in Individuals With Metabolic Syndrome
Brief Title: Periodized Aerobic Interval Training in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Laís M. Vanzella, Master Degree Student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53117116000005402
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Syndrome; Metabolic Syndrome X
Keywords: Metabolic syndrome X; Autonomic nervous system; Aerobic exercise; Exercise; Heart rate
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodized aerobic interval training (Experimental): The experimental groups will participate in a 16 week, three times a week based-program of periodized aerobic interval training that consist in warming [5 minutes of general stretching and 5 minutes of walking on treadmill with heart rate less than 20 percent of heart rate reserve (HHR)], followed by periodized aerobic interval training on treadmill, and cooling down [5 minutes of walk in treadmill with a heart rate less than 20 percent of HRR and 5 minutes of rest]
  Interventions: Behavioral: Periodized aerobic interval training
- Control group (No Intervention): Participants in the control group will be instructed not to take part in any regular exercise programs during the study period.

INTERVENTIONS:
Behavioral: Periodized aerobic interval training — The periodized training program consist in 3 phases: light (I) (training range varying between 20 to 39% of heart rate reserve and active recuperation of 19% of heart rate reserve); moderate (II) (training range varying between 40 to 59% of heart rate reserve and active recuperation of 30% of heart rate reserve) and high (III) (training range varying between 70 to 90 % of heart rate reserve and active recuperation of 50% of heart rate reserve).
  Arms: Periodized aerobic interval training

SUMMARY:
Autonomic disfunction present in metabolic syndrome subjects is related by a greater vulnerability of the heart and risk of cardiovascular events. In this context, aerobic interval training has been highlighted by its easy applicability and benefits effects in autonomic modulation in different populations. Therefore the studies that use de aerobic interval training in this different populations didn't realize a periodization of training with preparatory periods with progressive increase of load, specific phases with less duration predominating the intensity and transition periods for recuperation. Additionally, there isn't studies that investigate the effects of aerobic interval training in autonomic modulation of individuals with metabolic syndrome. In this context, periodized aerobic interval training can arise like a new type of treatment that offering security and efficacy in subjects with metabolic syndrome. So, the aim of the study is evaluate the effect of periodized aerobic interval training in cardiac autonomic modulation and cardiovascular and anthropometric parameters of individuals with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome according to international diabetes federation (IDF) definition
* Aged between 40 to 60 years

Exclusion Criteria:

* Participants who are currently participating in any regular exercise programs last six months;
* Use of drugs or medication (Except for risk factors of metabolic syndrome control);
* Inflammatory or infectious process;
* Musculotendinous or osteoarticular injuries in the lower limbs and/or spine;
* Chronic pulmonary disease;
* Neurological disorders;
* Cardiovascular disease.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 16 week after allocation

SECONDARY OUTCOMES:
Cardiovascular parameter : heart rate | 16 week after allocation
Cardiovascular parameter: blood pressure | 16 week after allocation
Anthropometric parameter: hit waist ratio | 16 week after allocation
Anthropometric parameter: abdominal circumference | 16 week after allocation
Anthropometric parameter: body mass index | 16 week after allocation
  Measured by weight and height

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, PHD, Study Director — Universidade Estadual Paulista - UNESP campus de Presidente Prudente
Locations (1):
- Laís Manata Vanzella, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
I don't have plans

REFERENCES:
- [Derived] Vanzella LM, Linares SN, Miranda RAT, Silva AKFD, Christofaro DGD, Netto Junior J, Vanderlei LCM. Effects of a new approach of aerobic interval training on cardiac autonomic modulation and cardiovascular parameters of metabolic syndrome subjects. Arch Endocrinol Metab. 2019 Mar-Apr;63(2):148-156. doi: 10.20945/2359-3997000000111. Epub 2019 Mar 21. PMID 30916161